CLINICAL TRIAL: NCT05974371
Title: A Basic Science Study on Episodic Memory Integration and Interference in Healthy Adults
Brief Title: Episodic Memory Integration and Interference
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston College (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: MH134570
Record Dates: First submitted 2023-07-26; First posted 2023-08-03 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-07

CONDITIONS: Episodic Memory

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Emotional memory updating paradigm (Experimental): All participants will encode AB/AC word pairs shown with images that have differing emotional valence (positive, negative, or neutral)
  Interventions: Other: emotional context similarity

INTERVENTIONS:
Other: emotional context similarity — On Day 1, all participants will encode AB neutral word pairs (e.g., Pencil - Car) shown with positive, negative, or neutral images. On Day 2, all participants will encode AC neutral words pairs (e.g., Pencil - Book) alongside images of either the same or different valence. The emotional similarity of AB (Day 1) and AC (Day 2) image contexts (i.e., the independent variable) will consist of the following conditions: positive-positive, positive-negative, negative-negative, negative-positive, neutral-neutral, neutral-positive, and neutral-negative.

SUMMARY:
The purpose of this study is to assess how emotional memories integrate and interfere with one another over time. We will be using a multi-session experimental paradigm consisting of two encoding sessions and one retrieval session. Participants will either complete these sessions online or in-person, with the latter collecting functional magnetic resonance imaging during the two encoding sessions.

DETAILED DESCRIPTION:
After being informed about the study, all participants giving written informed consent will complete three experimental sessions. On Day 1, participants will encode AB neutral word pairs (e.g., Pencil - Car) shown alongside positive, negative, or neutral images. Participants will also rate the images on valence and arousal. After encoding all stimuli, participants will immediately complete a retrieval task, during which they will be presented with the cue word (A; e.g., Pencil) and asked to recall the corresponding associate (B, e.g., Car). If incorrect, the correct word pair will be shown before the next trial. The complete list of word pairs will be shown until at least 90% of the word associates are recalled. On Day 2 (~24 h later), participants will return to encode new AC word pairs, where one of the words is the same from the first encoding session and one is different (e.g., Pencil - Book). These AC words pairs will be encoded alongside new images that either match the valence of the first session or shift to a different valence. Again, participants will rate the valence and arousal of each image and complete a subsequent memory test until they reach 90% accuracy on all word pairs. On Day 3, participants will complete the final session of the study, during which they will be shown a cue word (e.g., Pencil) and asked to freely recall the corresponding associates from days 1 and 2 (e.g., Car and Book). Participants will also be asked to remember the day each word associate was originally shown and the valence of the paired image from that day. 100 participants will complete these sessions and their corresponding behavioral tasks online (e.g., via Prolific). An additional 50 participants will complete these sessions in-person, and functional magnetic resonance imaging will be collected during Day 1 and Day 2 to examine how the blood oxygen-level dependent (BOLD) signal is modulated by task conditions. Psychophysiological data such as respiration and heart rate may also be collected. All participants (online and fMRI) will provide individual difference metrics on mood and well-being, including the Beck Depression Inventory, State-Trait Anxiety Inventory, NEO Personality Inventory, and Ruminative Responses Scale. On each day prior to the start of the experimental task, participants will also complete the Profile of Mood States, Positive and Negative Affect Scale, the Pittsburgh Sleep Quality Index, and sleep logs for the night before to index the amount and quality of sleep.

ELIGIBILITY:
Inclusion Criteria:

1. All participants: willing and able to follow the protocol
2. All participants: fluent in English
3. Online participants: online account in the crowdsourcing platform that will be used (e.g., Prolific)

Exclusion Criteria:

1. All participants: history of a psychiatric or neurological condition, and/or current psychotropic drug use (indicated by the participant)
2. fMRI participants: pregnant, metal in body (incl piercings or metallic makeup if unwilling to remove), unable to lie still for duration of scan (e.g., due to pain), Meniere's disease, claustrophobic, or other contraindication for MRI as determined my MRI technician, left-handed

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Memory for the Associated Words | Day 3
  During the memory recall task on Day 3, participants will be shown a cue word (A) and asked to recall the corresponding associates from Day 1 (B) and Day 2 (C) by typing their response in a blank text field. Participants will also report their confidence in these memories from 1 (not at all confident) to 9 (extremely confident).
fMRI Measured Neural Reactivity (Blood Oxygen-Level Dependent Signal) | Day 2
  fMRI data from Day 1 and Day 2 will be used to perform whole-brain analyses of neural response during encoding, as well as compute neural pattern similarity scores between AB and AC pairs from same- or differently-valenced contexts. Our primary hypothesis is that the similarity of neural patterns in the dorsomedial prefrontal cortex will predict memory performance on Day 3.

SECONDARY OUTCOMES:
Source Memory | Day 3
  During the memory recall task on Day 3, participants will also be asked to report which day each paired associate (B & C) was shown by selecting "1", "2", or "?" if unsure. Additionally, participants will indicate the valence of the image that they remember being associated with each pair from 1 (very negative) to 9 (very positive), as well as their confidence in the remembered valence from 1 (not at all confident) to 9 (extremely confident).
Change in Resting-State Functional Connectivity | Day 2
  Prior work from our lab has shown that increased amygdala-visuosensory connectivity after encoding predicts a memory bias for negatively-valenced stimuli, whereas increased amygdala-prefrontal connectivity predicts a memory bias for positively-valenced stimuli. In the current study, we will also examine whether changes in functional connectivity of the amygdala on Day 2 predict individual differences in memory performance on Day 3 (change = post - pre connectivity strength).

CONTACTS AND LOCATIONS:
Locations (1):
- Boston College, Chestnut Hill, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: De-identified data will be available for access and sharing as soon as the final version of the manuscript is accepted for publication
Access Criteria: Because data will be de-identified, these data will be posted on an open access website.